CLINICAL TRIAL: NCT03815279
Title: Iceland Screens Treats or Prevents Multiple Myeloma (iStopMM): A Nationwide Phase 2 Trial of Patients With Smoldering and Active Multiple Myeloma (MM)
Brief Title: A Nationwide Phase 2 Trial of Patients With Smoldering and Active Multiple Myeloma (MM)
Acronym: iStopMM
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Landspitali University Hospital (Other)
Collaborators: Amgen (Industry); Celgene (Industry); University of Iceland (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSH-17-001
Record Dates: First submitted 2019-01-09; First posted 2019-01-24 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma
Keywords: Multiple Myeloma; Smoldering Multiple Myeloma; Carfilzomib; Lenalidomide; Screening
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: An investigator initiated, academic, non-randomized, open-label phase 2 study that will assess carfilzomib, lenalidomide and dexamethasone regimen as treatment in patients with intermediate-risk (not carfilzomib) or high-risk SMM or active MM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-risk SMM and MM (Experimental): Twelve cycles of Carfilzomib-Lenalidomide-Dexamethason. Each cycle is 28 days. Carfilzomib intravenous, days 1, 8 and 15 (starting dose, 20 mg/m2 on day 1 of cycle 1; target dose, 56 mg/m2 thereafter) during cycles 1 through 12.
  Lenalidomide 25 mg orally once a day (3 weeks on/one week off) for 52 weeks. Dexamethasone 40 mg weekly for 16 weeks then 20 mg weekly for 16 weeks and thereafter 10 mg weekly for 16 weeks.
  Maintenance (1 year):
  Carfilzomib intravenous days 1 and 15 (56 mg/m2) during cycles 13 through 24. Lenalidomide 10 mg orally once a day (3 weeks on/one week off) for 52 weeks Dexamethasone 10 mg weekly for 52 weeks.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- Intermediate-risk SMM (Experimental): Lenalidomide 25 mg orally once a day (3 weeks on/one week off) for 52 weeks. Dexamethasone 40 mg weekly for 16 weeks, then 20 mg weekly for 16 weeks.
  Maintenance (1 year):
  Lenalidomide 10 mg orally once a day (3 weeks on/one week off) for 52 weeks.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be administered intravenously three times per cycle (28 day cycles) for cycle 1-12. Thereafter twice per cycle for cycle 13-24
  Other Names: Kyprolis
  Arms: High-risk SMM and MM
Drug: Lenalidomide — Lenalidomide PO once daily on days 1-21 of a 28 day cycle
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone will be administered weekly
  Other Names: Dexasone

SUMMARY:
The purpose of this study is to determine the efficacy of treating patients with intermediate risk smoldering multiple myeloma (SMM) with combinational therapy with dexamethasone and lenalidomide (Rd) and patients with high risk SMM with combinational therapy with Rd and carfilzomib.

DETAILED DESCRIPTION:
This is an open label, single center, phase II study assessing the efficacy of treating patients with intermediate-risk smoldering myeloma (SMM) with combinational therapy with dexamethasone and lenalidomide and treating patients with high risk SMM and active multiple myeloma (MM) with combinational therapy with dexamethasone, lenalidomide and carfilzomib. Patients that are eligible for this study are participants in the IstopMM study (ClinicalTrials.gov number, NCT03327597) that are diagnosed with intermediate or high-risk SMM or active MM.

ELIGIBILITY:
Inclusion Criteria:

Participants that are diagnosed with MM, high- or intermediate-risk SMM in the iStopMM study will be invited to participate in this study. Each patient must meet all the following inclusion criteria to be enrolled in the study:

1. Age more than 18 years.
2. Active MM or
3. Smoldering myeloma, which is untreated, as defined by: Measurable M spike OR pathological FLC ratio AND bone marrow PC% > 10%
4. The following laboratory values obtained ≤ 30 days prior to registration

   * Calculated creatinine clearance ≥ 30mL/min (using CKD-EPI equation)
   * Absolute neutrophil count (ANC) > 1000/mm3
   * Platelet count > 75000/mm3
   * Hemoglobin ≥ 8.0 g/dL
   * Total bilirubin ≤ 1.5 x ULN
   * ALT and AST ≤ 3 x ULN
5. Measurable disease as defined by at least one of the following:

   * Serum monoclonal protein > 1.0g/L
   * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
   * Serum immunoglobulin free light chain ≥ 10 mg/dL and abnormal serum immunoglobulin kappa to lambda free light chain ratio
6. Prior therapy for the treatment of solitary plasmacytoma is permitted, but >7 days should have elapsed from the last day of radiation. NOTE: Prior therapy with clarithromycin, DHEA, anakinra, pamidronate or zoledronic acid is permitted. Any additional agents not listed must be approved by the Principal Investigator.
7. ECOG performance status 0, 1 or 2
8. Negative pregnancy test done ≤7 days prior to C1D1, for women of childbearing potential only.
9. Willing to follow strict birth control measures as outlined in the protocol.
10. Female subjects: If they are of childbearing potential, agree to one of the following:

    Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of trial drug, AND must also adhere to the guidelines of any treatment-specific pregnancy prevention program (appendix 1), if applicable, OR Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
11. Male subjects: even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following: Agree to practice effective barrier contraception during the entire trial treatment period and through 90 days after the last dose of trial drug, OR Must also adhere to the guidelines of any treatment-specific pregnancy prevention program (appendix 1), if applicable, OR Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). Willing to return to enrolling institution for follow-up during the Active Treatment Phase of the trial. Agree not to donate sperm for at least 90 days after the last dose of carfilzomib
12. Willing to provide samples for planned research
13. Life expectancy > 6 months

Exclusion Criteria:

1. MGUS or low-risk smoldering myeloma.
2. Diagnosed or treated for another malignancy ≤ 2 years before trial enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. NOTE: Subjects with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
3. If any of the following exist at screening, subject will not be eligible for trial because this trial involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown: Pregnant women Nursing women Men or women of childbearing potential who are unwilling to employ adequate contraception (per protocol)
4. Other co-morbidity which would interfere with subject's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
5. Other concurrent chemotherapy, or any ancillary therapy considered investigational.

   NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment.
6. Peripheral neuropathy > Grade 3 on clinical examination or grade 2 with pain within 30 days prior to C1D1.
7. Major surgery ≤14 days prior to C1D1.
8. Evidence of current uncontrolled cardiovascular conditions, including hypertension, cardiac arrhythmias, congestive heart failure, unstable angina, or myocardial infarction within the past 6 months. Note: Prior to trial entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
9. Known human immunodeficiency virus (HIV) positive.
10. Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
11. Any medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
12. Known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or Investigator's Brochure), or known sensitivity to mammalian-derived products.

    Known allergies, hypersensitivity, or intolerance to trial drugs.
13. Inability to comply with protocol/procedures.
14. LVEF < 40% for patients treated with carfilzomib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD negativity | 36 months after study enrollment
  Minimal residual disease (MRD) as determined VDJ sequencing

SECONDARY OUTCOMES:
Progression free survival | Up until 3 years after treatment
  Rates of progression free survival with progression being determined by IMWG response criteria
Overall survival | Up until 3 years after treatment
  Overall survival as determened by the Icelandic National Cause of Death Registry

CONTACTS AND LOCATIONS:
Overall Officials: Sigurdur Y Kristinsson, MD, PhD, Principal Investigator — Landspitali University Hospital
Locations (1):
- Landspitali University Hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No